CLINICAL TRIAL: NCT00470132
Title: Ventricular Shunt and Drain Infections - Timing of Reimplantation
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO07040262
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Ventricular Shunt Infection
Keywords: ventricular shunt

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The retrospective study will help determine whether or not placement of new devices prior to the recommended time was associated with a high risk of relapse or treatment failure.

DETAILED DESCRIPTION:
The following information will be collected from the medical record retrospectively: demographic data (age, gender, ethnicity, height, weight), past medical history, laboratory results, microbiologic data, data on the patients' devices (type of device, data that it was placed, exchanged or removed), treatment and clinical and microbiological outcomes. This will all be collected retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients that were cared for by the PI for the purpose of treating an infected ventricular shunt or drainage device for the central nervous system.

Exclusion Criteria:

* Those patients records that do not meet entry criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: infected ventricular shunt
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Byers, MD, Principal Investigator — University of PIttsburgh and UPMC
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States